CLINICAL TRIAL: NCT01869829
Title: International Pediatric Fungal Network: Multi-Center Studies to Improve Diagnosis and Treatment of Pediatric Candidiasis
Brief Title: PEACE: Pediatric Antifungal Comparative Effectiveness
Acronym: PEACE
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Children's Hospital of Philadelphia (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00045657; 1R01AI103315-01A1 (NIH)
Record Dates: First submitted 2013-05-31; First posted 2013-06-05 (Estimated); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Pediatric Invasive Candidiasis
Keywords: Candida; Pediatric; Antifungal
MeSH Terms: conditions — Torulopsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Weeks
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Pediatric Invasive Candidiasis: Pediatric patients (age > 120 days and < 18 years) with documented proven or probable invasive candidiasis
  Interventions: Drug: Observational antifungal therapy

INTERVENTIONS:
Drug: Observational antifungal therapy — Observational study of primary antifungal therapy utilized and outcomes, including:
  fluconazole, voriconazole, amphotericin B, caspofungin, and micafungin
  All agents are given as standard of care.

SUMMARY:
The overarching objective is to develop new evidence-based treatment guidelines for invasive fungal diseases in children. To accomplish that, this protocol will focus on two specific aims: 1) Compare the effectiveness of echinocandin versus amphotericin B or triazole antifungal therapy for pediatric invasive candidiasis and for the subset of patients with invasive candidemia; 2) Characterize the incidence rate of inpatient pediatric invasive candidiasis per hospital admissions.

DETAILED DESCRIPTION:
This study is a multicenter, national and international, prospective observational comparative effectiveness study.

The primary aim of this study is to compare the effectiveness of echinocandin versus amphotericin B or triazole antifungal therapy for pediatric invasive candidiasis and for invasive candidemia. The primary effectiveness endpoint for study aim 1 is the comparison of global response at 14 days of antifungal therapy between antifungal therapeutic classes. The secondary effectiveness endpoints for study aim 1 are comparative effectiveness of the 1) global response to antifungal therapy after 30 days and 2) all-cause mortality at 30 days.

The secondary aim is to characterize the frequency of pediatric candidiasis by describing the incidence of pediatric candidiasis relative to all pediatric admissions. For this aim, the investigators will use descriptive statistics to establish the frequency of hospital admissions involving an invasive candidiasis per total hospital admissions and total hospital days during the study period.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females age > 120 days and <18 years
2. Documented proven or probable case of invasive candidiasis
3. Parental/guardian permission (informed consent, if required) and if appropriate, child assent (if required).

Exclusion Criteria:

1) Any history of prior Candida infection within the previous 35 days (These patients will not be eligible for analysis in aim 1 but will be eligible for inclusion of aim 2)

Ages: 120 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients with invasive candidiasis
Sampling Method: Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2015-01; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Global response to antifungal therapy | 14 days

SECONDARY OUTCOMES:
Global response of antifungal therapy | 30 days
All-cause mortality | 30 days

OTHER OUTCOMES:
Incidence of pediatric invasive fungal infections | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: William J Steinbach, MD, Principal Investigator — Duke University; Theoklis E Zaoutis, MD MSCE, Principal Investigator — Children's Hospital of Philadelphia
Locations (35):
- United States (27):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital at Stanford, Palo Alto, California
  - Rady Children's Hospital, San Diego, California
  - UCSF Benioff Children's Hospital, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - All Children's Hospital, St. Petersburg, Florida
  - Ann and Robert Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital and Clinics of Minnesota, Minneapolis, Minnesota
  - Children's Mercy, Kansas City, Missouri
  - Cohen Children's Medical Center of New York, New Hyde Park, New York
  - New York Presbyterian Phyllis and David Komansky Center for Children's Health, New York, New York
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Children's, Cleveland, Ohio
  - OHSU Doernbecher Children's Hospital, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee
  - Dell Children's Medical Center, Austin, Texas
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- The Hospital for Sick Children, Toronto, Canada
- Colombia (2):
  - Centro de Estudios en Infectologia Pediatricia, Cali
  - Centro Medico Imbanaco, Cali
- 3rd Department Pediatrics Aristole University School of Medicine, Hippokration Hospital, Thessaloniki, Greece
- Postgraduate Institute of Medical Education and Research, Chandigarh, India
- Instuto Giannina Gaslini, Genoa, Italy
- King Faisal Specialist Hospital & Research Center, Riyadh, Saudi Arabia
- Hospital d'Universitari Vall d'Hebron, Barcelona, Spain

REFERENCES:
- [Result] Fisher BT, Zaoutis TE, Xiao R, Wattier RL, Castagnola E, Pana ZD, Fullenkamp A, Boge CLK, Ross RK, Yildirim I, Palazzi DL, Danziger-Isakov L, Vora SB, Arrieta A, Yin DE, Aviles-Robles M, Sharma T, Tribble AC, Maron G, Berman D, Green M, Sung L, Romero J, Hauger SB, Roilides E, Belani K, Nolt D, Soler-Palacin P, Lopez-Medina E, Muller WJ, Halasa N, Dulek D, Hussain IZB, Pong A, Hoffman J, Rajan S, Gonzalez BE, Hanisch B, Aftandilian C, Carlesse F, Abzug MJ, Huppler AR, Salvatore CM, Ardura MI, Chakrabarti A, Santolaya ME, Localio AR, Steinbach WJ. Comparative Effectiveness of Echinocandins vs Triazoles or Amphotericin B Formulations as Initial Directed Therapy for Invasive Candidiasis in Children and Adolescents. J Pediatric Infect Dis Soc. 2021 Aug 10:piab024. doi: 10.1093/jpids/piab024. Online ahead of print. PMID 34374424
- See also: International Pediatric Fungal Network — http://www.ipfn.org/